CLINICAL TRIAL: NCT03075813
Title: Early Recognition and Response to Increases in Surgical Site Infections Using Optimized Statistical Process Control Charts
Brief Title: Early Recognition and Response to Increases in Surgical Site Infections Using Optimized Statistical Process Control Charts: The Early 2RIS Study
Acronym: Early 2RIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00081013
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Infection Control; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Cluster (Experimental): Surgical surveillance data submitted to the DICON Surgical Database will undergo immediate analysis by optimized SPC methods. If a signal is generated, study personnel in DICON will be notified to adjudicate the signal and determine if further action is required.
  Optimized SPC methods include the application of two SPC charts. The investigator determined that when either chart identifies a signal, the study will have approximately 90% sensitivity and 65% specificity to identify important increases in rates of SSI.
  Interventions: Other: Intervention Cluster
- Control Cluster (No Intervention): Local personnel in clusters randomized to traditional surveillance and feedback will receive bar graph reports and data interpretation per routine DICON surveillance. These reports will be provided every 6 months.

INTERVENTIONS:
Other: Intervention Cluster — Surgical surveillance date will be analyzed by optimized SPC methods. if signal is generated, study personnel in DICON will be notified to adjudicate the signal and determine if further action is needed.
  Arms: Intervention Cluster

SUMMARY:
The purpose of this quality improvement study is to measure the effectiveness of surveillance using optimized statistical process control (SPC) methods and feedback on rates of surgical site infection (SSI) compared to traditional surveillance and feedback.

The primary objective is to determine if hospital clusters randomized to receive feedback from optimized SPC surveillance methods collectively have lower rates of SSI compared to hospital clusters randomized to receiving feedback from traditional surveillance methods. Secondary objectives are 1) to estimate and compare the number of signals identified using optimized SPC methods and traditional surveillance methods; 2) to estimate and compare the time and effort required to investigate signals generated using optimized SPC methods and traditional surveillance methods; and 3) to estimate the number and proportion of false-positive signals identified using optimized SPC methods and traditional surveillance methods.

The Early 2RIS study will be a prospective, multicenter cluster randomized controlled trial using stepped wedge design. The active component of the quality improvement study will be performed in 29 DICON hospitals over three years, from March 2017 through February 2020. Clusters randomized to intervention will receive feedback on increasing rates of SSI identified through optimized SPC methods. This intervention is expected to decrease the subsequent rate of SSIs by closing the feedback loop on SSI outcomes.

Participating study hospitals will all be members of DICON, a network of 43 community hospitals in North Carolina, South Carolina, Georgia, Florida, and Virginia that provides community hospitals access to consultative services from infection prevention experts, data analyses and benchmarking, and educational materials designed by faculty from Duke. This study is considered part of routine quality improvement measures and a part of previously established agreements between DICON and the community hospitals. Data flow and communication are outlined in detail in approved protocols determined to be exempt research by the DUHS IRB. Briefly, existing clinical data are extracted from participating hospitals' electronic medical record into discrete files according to DICON specifications. Then a de-identification process removes direct patient identifiers into a limited dataset.

The majority of data collection will occur through methods already developed and utilized by study hospitals. In brief, each hospital routinely submits limited datasets to the DICON Surgical Surveillance Database, including the following variables: hospital, type of procedure, patient identifier, date of procedure, age, sex, surgeon identifier, start/stop times, ASA score, wound class, risk index, SSI (Yes/No), date of infection, type of SSI, location at diagnosis and organism. No identifiable patient or surgeon data are transmitted to the DICON Surgical Database. Data definitions and data collection methods are standardized across DICON hospitals. Following signal adjudication, additional data will be collected in a REDCap database to document actions and rationale.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo one of 13 targeted procedures in 29 DICON study hospitals will be eligible for inclusion. The 13 targeted procedures include coronary artery bypass graft, cardiac valve replacement, colon surgery, herniorrhapy, knee arthroplasty, hip arthroplasty, Cesarean section, abdominal hysterectomy, vaginal hysterectomy, spinal fusion, laminectomy, carotid endarterectomy, and peripheral venous bypass. These procedures were selected because they are frequently performed in community hospitals and/or are associated with particularly adverse outcomes if complicated by SSI. Eligible procedures will be categorized by procedure type at each hospital using ICD9 codes published by the NHSN, per routine DICON activities. Six clusters were constructed from these procedures to ensure that surgeons who perform similar types of procedures were grouped together to limit potential bias. These clusters are labeled as Spine, GI, OB/GYN, Ortho, Vascular, and Cardiac. These clusters are the units for randomization and analysis.

Exclusion Criteria:

* DICON hospitals that did not submit a letter of support for participating in the study will be excluded. Patients not undergoing one of these 13 procedure types at the 29 study hospitals will be excluded from the analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Differences in rates of SSI. | SSIs can be diagnosed up 30 to 90 days following the procedure, depending on the type of procedure
  SSI rate will be calculated as number of SSI/100 procedures per month
  SSIs will be defined using standard NHSN definitions
  DICON personnel train local infection preventionists about how to use and interpret SSI definitions. Thus, standard definitions and methods are used at all study hospitals.
  Cluster-level risk adjustment will be performed using median surgical volume and median NHSN Risk Index (an operation- and patient-specific risk score that predicts SSI) per cluster.

SECONDARY OUTCOMES:
Proportion of SSIs determined to be potentially preventable | diagnosed up 30 to 90 days following the procedure, depending on the type of procedure
  Among SSIs investigated, each will be provided a "preventability score" after reviewing if best practices were followed.
Description of and difference in number and type of signals | 36 months (entire study period)
  Signals identified using optimized SPC will be compared to signals identified using standard surveillance; Not a patient-specific outcome
Difference in number of outbreaks identified | 36 months (entire study period)
  Outbreaks identified using optimized SPC will be compared to outbreaks identified using standard surveillance; Not a patient-specific outcome
Difference in number of investigations of increased rates of SSI | 36 months (entire study period)
  Signals may or may not lead to subsequent investigation. Investigators will compare the number of investigations performed following the use of optimized SPC to the number of investigations performed following the use of standard surveillance; signals identified using standard surveillance; Not a patient-specific outcome
Total number and differences in proportion of signals that led to investigations | 36 months (entire study period)
  Signals may or may not lead to subsequent investigation. Investigators will compare the number of investigations performed following the use of optimized SPC to the number of investigations performed following the use of standard surveillance; signals identified using standard surveillance; Not a patient-specific outcome
Time required to investigate signals | 36 months (entire study period)
  Investigators will monitor the time required to investigate signals and compare the time required following the use of optimized SPC methods to the time required following the use of standard surveillance; not a patient-specific outcome
Timing of signals | 36 months (entire study period)
  Investigators will determine how promptly the different surveillance strategies identify signals and compare average/median time to signal between the two study arms; not a patient-specific outcome
Time to completion of investigation | 36 months (entire study period)
  Investigators will determine the time required to complete investigations
Strength and type of signals | 36 months (entire study period)
  Investigators will compare the strength and types of signals generated from each type of surveillance with subsequent adjudication and intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Deverick Anderson, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baker AW, Ilies I, Benneyan JC, Lokhnygina Y, Foy KR, Lewis SS, Wood B, Baker E, Crane L, Crawford KL, Cromer AL, Padgette P, Roach L, Adcock L, Nehls N, Salem J, Bratzler D, Dellinger EP, Greene LR, Huang SS, Mantyh CR, Anderson DJ. Early recognition and response to increases in surgical site infections using optimised statistical process control charts-The early 2RIS trial: A multicentre stepped wedge cluster randomised controlled trial. EClinicalMedicine. 2022 Oct 17;54:101698. doi: 10.1016/j.eclinm.2022.101698. eCollection 2022 Dec. PMID 36277312
- [Derived] Anderson DJ, Ilies I, Foy K, Nehls N, Benneyan JC, Lokhnygina Y, Baker AW. Early recognition and response to increases in surgical site infections using optimized statistical process control charts-the Early 2RIS Trial: a multicenter cluster randomized controlled trial with stepped wedge design. Trials. 2020 Oct 28;21(1):894. doi: 10.1186/s13063-020-04802-4. PMID 33115527